CLINICAL TRIAL: NCT02847676
Title: Differences in Peritoneal Stem Cells in Women With and Without Adhesions After Gynaecological Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pius-Hospital Oldenburg (Other)
Collaborators: University of Leipzig (Other); University of Oldenburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. med. Rudy Leon De Wilde, Prof. Dr. Dr. med, Pius-Hospital Oldenburg
Other Study IDs: PHDW-005
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Peritoneal Adhesions
Keywords: Peritoneal adhesions; Stem cells; MSC

STUDY DESIGN:
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Peritoneal tissue samples taken from Adhesions, Peritoneal lining and omentum.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- No previous surgery, adhesions present.: Patients have had no previous abdominal surgery. Inspection shows peritoneal adhesions.
  Interventions: Procedure: Tissue sample donation
- No previous surgery, no adhesions present.: Patients have had no previous abdominal surgery. Inspection shows no peritoneal adhesions.
  Interventions: Procedure: Tissue sample donation
- Previous surgery, adhesions present.: Patients have had previous abdominal surgery. Inspection shows peritoneal adhesions.
  Interventions: Procedure: Tissue sample donation
- Previous surgery, no adhesions present.: Patients have had previous abdominal surgery. Inspection shows no peritoneal adhesions.
  Interventions: Procedure: Tissue sample donation

INTERVENTIONS:
Procedure: Tissue sample donation — Patients undergo planned gynaecological surgery. Tissue samples, which are routinely taken, are donated.

SUMMARY:
Our study aims to characterise a possible pluripotent cell population in the abdomen responsible for peritoneal adhesions. We therefore want to take samples from women undergoing planned laparoscopic surgery with and without adhesions, isolate the cells and characterise them for markers of pluripotency.

DETAILED DESCRIPTION:
Peritoneal adhesions are connective tissue bands between two normally separate anatomical structures within the abdominal or pelvic cavity. Those adhesions can occur after gynaecological or other surgeries involving the pelvis or abdomen. Adhesions have severe clinical as well as economical Consequences. There is substantial morbidity (from chronical pain to obstructions and infertility) and a higher surgical risk if additional surgery is needed, due to a higher intraoperative blood loss and a higher incidence of lacerations when peritoneal adhesions are present. In combination with a prolonged surgery duration, the economical impact is tremendous. A 2011 study estimated the cost of adhesion - related surgeries to be 2,3 billion US dollar exclusively in the USA. 46.3% of those surgeries had their origin or localisation in the gynaecological area. The genesis of adhesiolysis - obligatory peritoneal adhesions remains unclear to this date.

After all surgeries cytokine induced fibrotic bands appear within 72 hours. Usually those bands are eliminated by a fibrinolytic sequence within 10 days.

For Adhesions that persist afterwards the generally accepted assumption is, that there is a failure of the fibrinolytic sequence with unknown origin. Adhesions which persist for more than 10-14 days become thicker and vascularised. In those "adult" adhesions not only fibrin is found but also fat tissue, smooth muscles and myelinised and un - myelinised axons.

In developmental biology those tissues differentiate from different germ layers, namely mesoderm and ectoderm. Finding cells from multiple germ layers points towards a pluri -, multi-, or stem cell like precursor cell from which those adhesions develop. Such a cellpopulation has not been characterised in the abdomen to the date of writing, though Studies have shown evidence (ranging from mesothelial - to - mesenchymal shift to Clusters of differentiation from multiple germ layers) which made multiple researchers postulate a pluripotent precursor cell located in the submesothelium.

In our research we will therefore take peritoneal samples from adhesions, peritoneal wall lining and omentum in subjects with and without peritoneal adhesions in subjects undergoing indicated laparoscopic surgery at the gynaecological ward at the Pius hospital in Oldenburg.

The samples are routinely taken as part of the procedure and usually discarded. At least 24 hours prior to surgery, the subjects will have a chance to give their informed consent to donate those samples for our study. The study is thus designed in a way that subjects won't undergo additional risk by participating in the study. Taking part or the refusal hereof won't have any effect on the treatment or surgical outcome for the subjects. Also, taking part in our study won't have any benefits or additional risks for the subjects.

The samples will then be taken to the university of Leipzig, where we will culture, isolate and characterise the cells. Characterisation will mostly be the application of pluripotency markers, cell sorting and immunoassays. Expression profiles will be used to further understand the mesothelial - to - mesenchymal shift. Depending on our findings the protocol for analysis will be adjusted in consultation with Prof. dr. dr. De Wilde and Prof. dr. Bader.

The study will approximately take 6 months, with an additional 6 months for writing and publication. The study is funded by the research funding pool of the university of Oldenburg.

ELIGIBILITY:
Inclusion Criteria:

1. Woman equal to and above 18 years of age.
2. Woman with a negative pregnancy test at the time of recruitment, and sufficient contraception from time of
3. Woman with any gynecological pathology requiring scheduled pelvic gynecological surgery, either laparotomy or laparoscopy.
4. Woman without primary peritoneal disease.

Exclusion Criteria:

1. Woman with a primary peritoneal pathology.
2. Emergency surgery
3. Patients under systemic immunosuppressive therapy in the previous 6 months
4. Patients with current intra-abdominal or pelvic abscess or systemic infection
5. Pregnant woman
6. Simultaneous participation in another clinical trail

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing scheduled pelvic gynecological surgical treatment, at the Gynecology Department of Pius Hospital, Oldenburg.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pluripotency markers (Sox2, Nanog, Klf 4, Oct 3/4) | at least 10
  days since previous surgery

IPD SHARING:
Plan to Share IPD: No